CLINICAL TRIAL: NCT01718028
Title: The Effect of SYSTANE® BALANCE on Non-Invasive Tear Film Break Up Time (NITFBUT) in Dry Eye Subjects With Lipid Deficiency Following 30 Days of Use
Brief Title: The Effect of SYSTANE® BALANCE on Tear Film Break Up Time in Dry Eye Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDG-11-262
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Dry Eye
Keywords: Systane BALANCE; Dry eye; lipid deficiency; NITFBUT
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Propylene Glycol; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYSTANE® BALANCE (Experimental): Propylene glycol 0.6% ocular emulsion, 1 drop in each eye 4 times a day for 30 days
  Interventions: Other: Propylene glycol 0.6% ocular emulsion
- LARMABAK® (Active Comparator): Sodium chloride 0.9% saline solution, 1 drop in each eye 4 times a day for 30 days
  Interventions: Other: Sodium chloride 0.9% saline solution

INTERVENTIONS:
Other: Propylene glycol 0.6% ocular emulsion
  Other Names: SYSTANE® BALANCE
  Arms: SYSTANE® BALANCE
Other: Sodium chloride 0.9% saline solution
  Other Names: LARMABAK®
  Arms: LARMABAK®

SUMMARY:
The purpose of this study was to evaluate the ability of SYSTANE® BALANCE dosed 4 times a day for 30 days to increase non-invasive tear film break up time over baseline, compared to a saline control, in dry eye subjects with lipid deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Read, sign, and date an information consent;
* Willing and able to follow instructions and maintain the appointment schedule;
* Best-corrected visual acuity of 0.6 logMAR or better in each eye as assessed at Visit 1;
* Must not have used any topical ocular drops for approximately 24 hours prior to Visit 1;
* Meet protocol-specified criteria for dry eye at Visit 1;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History or evidence of ocular or intraocular surgery or serious ocular trauma in either eye within the past six months;
* Current punctal occlusion of any type (e.g., collagen plugs, silicon plugs);
* History of intolerance or hypersensitivity to any component of the study medications;
* History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia; active or recent varicella viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye;
* Use of any concomitant topical ocular medications during the study period;
* Use of systemic medications that may contribute to dry eye unless on a stable dosing regimen for a minimum of 30 days prior to Visit 1;
* Ocular conditions such as conjunctival infections, iritis, or any other ocular condition that may preclude the safe administration of either drop under investigation;
* Unwilling to discontinue contact lens wear during the study period. Contact lens wear must have been discontinued at least one week prior to Visit 1.
* Participation in an investigational drug or device study within 30 days of entering this study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Consultório Oftalmológico, Martínez, Buenos Aires, Argentina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in Argentina.
Pre-assignment Details: Of the 51 enrolled, 2 participants withdrew their consent prior to receiving treatment and were exited from the study. This reporting group includes all participants who received treatment.
Period: Overall Study
Arm/Group | SYSTANE® BALANCE | LARMABAK®
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SYSTANE® BALANCE | LARMABAK® | Total
Number analyzed (Participants) | 25 | 24 | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 45.52 (20.06) | 42.96 (17.71) | 44.27 (18.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  Argentina | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in NITFBUT at Day 30
Description: NITFBUT is defined as the time elapsed between eye opening after a blink and the appearance of the first break in the tear film, ie, dry area. NITFBUT was evaluated noninvasively with a Tearscope. One eye from each participant was chosen as the study eye, and only data for the study eye contributed to the analysis. A positive change value indicates an improvement in tear film stability, which may improve dry eye symptoms in dry eye sufferers.
Time Frame: Baseline (Day 0), Day 30
Population: Intent-to-treat: All randomized participants who received test product and attended at least one on-therapy study visit
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SYSTANE® BALANCE | LARMABAK®
Number analyzed (Participants) | 25 | 24
seconds | 2.83 (0.74) | 0.66 (0.55)

2. Secondary Outcome: Mean Change From Baseline in NITFBUT at Day 14
Description: as for outcome 1
Time Frame: Baseline (Day 0), Day 14
Population: Intent-to-treat: All randomized participants who received test product and attended at least one on-therapy study visit
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SYSTANE® BALANCE | LARMABAK®
Number analyzed (Participants) | 25 | 24
seconds | 1.98 (0.60) | 0.65 (0.77)

3. Secondary Outcome: Mean NITFBUT by Visit
Description: NITFBUT is defined as the time elapsed between eye opening after a blink and the appearance of the first break in the tear film, ie, dry area. NITFBUT was evaluated noninvasively with a Tearscope. One eye from each participant was chosen as the study eye, and only data for the study eye contributed to the analysis. A longer tear film break-up time indicates a more stable tear film, which may improve dry eye symptoms in dry eye sufferers.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: Intent-to-treat: All randomized participants who received test product and attended at least one on-therapy study visit
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SYSTANE® BALANCE | LARMABAK®
Number analyzed (Participants) | 25 | 24
seconds
  Baseline | 4.60 (0.69) | 4.93 (0.80)
  Day 14 | 6.58 (0.74) | 5.57 (0.93)
  Day 30 | 7.43 (0.51) | 5.59 (0.66)

4. Secondary Outcome: Percent Change From Baseline in NITFBUT by Visit
Description: NITFBUT is defined as the time elapsed between eye opening after a blink and the appearance of the first break in the tear film, ie, dry area. NITFBUT was evaluated noninvasively with a Tearscope. One eye from each participant was chosen as the study eye, and only data for the study eye contributed to the analysis. The percentage of participants with a lengthening in tear film break up time relative to baseline is reported. A positive value indicates an improvement in film stability, which may improve dry eye symptoms in dry eye sufferers.
Time Frame: Baseline (Day 0), Day 14, Day 30
Population: Intent-to-treat: All randomized participants who received test product and attended at least one on-therapy study visit
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SYSTANE® BALANCE | LARMABAK®
Number analyzed (Participants) | 25 | 24
percent change
  Percent Change from Baseline at Day 14 | 44.99 (19.46) | 14.35 (17.88)
  Percent Change from Baseline at Day 30 | 65.03 (28.41) | 15.06 (14.48)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (1 month, 3 days). An adverse event was defined as any untoward medical occurrence in a subject administered the test product, regardless of causal relationship.
Description: This reporting group includes all participants who received at least one dose of Systane® BALANCE or saline solution.
Arm/Group | SYSTANE® BALANCE | LARMABAK®
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.